CLINICAL TRIAL: NCT03618498
Title: Internal Limiting Membrane Flaps for Coexistent Macular Hole and Retinal Detachment in Eyes of Proliferative Diabetic Retinopathy
Brief Title: Internal Limiting Membrane Flaps for Coexistent Macular Hole and Retinal Detachment
Acronym: ILMFCMHRDPDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, San Ni Chen, medical doctor, Changhua Christian Hospital
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180314
Record Dates: First submitted 2018-07-23; First posted 2018-08-07 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Retinal Detachment
Keywords: macular hole; retinal detachment; PDR
MeSH Terms: conditions — Retinal Detachment; Retinal Perforations

STUDY DESIGN:
Intervention Model Description: A 25-gauged blunt-tipped needle connected with Viscoat® (Alcon laboratories, Fort Worth, TX, USA) containing syringe was placed within the macular hole just below the level of the macular hole. A small amount of Viscoat® was injected into and around the hole. An ICG solution (25 mg ICG in 15 ml 5% glucose-water solution, final concentration = 1.7 mg/ml) was then carefully applied around the macular hole within the arcade.Excessive ICG was immediately removed by suction. ILM at the parafoveal area was peeled in a circular fashion. Care was taken not to peel the ILM flap across the hole edge. If possible, at least 1.5 to 2 disc area of partially detached ILM around the hole was left in place with central part remained attached to the edge of the hole.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient accept surgery (Other): Proliferative diabetic retinopathy suffering from MH with RD who were treated with vitrectomy combined with inverted epiretinal ILM flap,inverted ILM flaps insertion techniques, or free ILM flaps.
  Interventions: Procedure: ILM flaps insertion techniques or free ILM flaps.

INTERVENTIONS:
Procedure: ILM flaps insertion techniques or free ILM flaps. — The ILM flap anchoring on the hole edge was inverted and covered the hole.Otherwise, temporal side ILM flap was used. However, if the risk of ILM flipping back was judged to be high, ILM insertion instead of ILM hole coverage was adopted.If the size of the ILM flaps was judged inadequate, the double ILM insertion technique was used, done by adding a piece of previously obtained free ILM flap on top of the inverted ILM tissue until they were securely in place.

SUMMARY:
Purpose: To evaluate the logical surgical approaches in closing macular holes in eyes of proliferative diabetic retinopathy with retinal detachment

DETAILED DESCRIPTION:
High MH closure rate can be achieved. Other than high myopia, MH with RD may appear in several conditions, such as severe vitreomacular traction, proliferative diabetic retinopathy (PDR).clinical charts were reviewed of patients of proliferative diabetic retinopathy suffering from MH with RD who were treated with vitrectomy combined with inverted epiretinal ILM flap,inverted ILM flaps insertion techniques, or free ILM flaps.Standard 3-port 23 or 25 gauged pars plana vitrectomy was performed. After core vitrectomy, anterior-posterior oriented tractions as well as all fibrovascular tissues were removed as thoroughly as possible.The patients were kept in a facedown position overnight and were allowed to take any positions except supine for approximately one week.Various surgical approaches utilizing in managing macular hole may effectively closing macular holes and reattach retina.

ELIGIBILITY:
Inclusion Criteria:

* Patients were proliferative diabetic retinopathy suffering from MH with RD.

Exclusion Criteria:

* Patients were not proliferative diabetic retinopathy suffering from MH with RD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Wilcoxon Sign-Rank test | Baseline, 12 months.
  A statistical comparison of average of two dependent samples

CONTACTS AND LOCATIONS:
Overall Officials: Chen San-Ni, MD, Study Director — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR